CLINICAL TRIAL: NCT05956093
Title: FAST HOC-FAPI PET for Staging of High-Grade Serous Ovarian Cancer .
Brief Title: 68Ga-FAPI PET/CT in the Staging of High-Grade Epithelial Ovarian Cancers: A Pilot Study
Acronym: FAST HOC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-5070.0
Record Dates: First submitted 2023-06-08; First posted 2023-07-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: High Grade Serous Ovarian Cancer (HGSOC)

STUDY DESIGN:
Intervention Model Description: * This study focuses on individuals who have been diagnosed or are suspected to have high-grade serous ovarian cancers (HGSOC).
  * They must have had a CT scan of their abdomen and pelvis within 6 weeks before enrolling in the study and be at clinical stage III or IV.
  * These individuals must also be considered for primary cytoreductive surgery or neoadjuvant chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- high-grade epithelial ovarian cancers. (Experimental): individuals who have been diagnosed or are suspected to have high-grade serous ovarian cancers (HGSOC). They must have had a CT scan of their abdomen and pelvis within 6 weeks before enrolling in the study and be at clinical stage III or IV.
  Interventions: Radiation: FAPI PET CT

INTERVENTIONS:
Radiation: FAPI PET CT — the utilization of Gallium 68 labelled Fibroblast Activation Protein Inhibitor (68Ga-FAPI) PET/CT to accurately stage high-grade epithelial ovarian cancers.

SUMMARY:
The investigator will use a technology called PET-CT that combines a Positron Emission Tomography (PET) scan with a computed tomography (CT) scan. This combined imaging test, where PET and CT data are gathered at one time, will be performed on an integrated PET-CT scanner located at Princess Margaret Cancer Centre.

The purpose of this study is to find out if the use of 68Ga-PNT6555 (FAPI) PET-CT will improve the assessment of disease extent as compared to routine CT scans.

DETAILED DESCRIPTION:
The investigator will use a technology called PET-CT that combines a Positron Emission Tomography (PET) scan with a computed tomography (CT) scan. This combined imaging test, where PET and CT data are gathered at one time, will be performed on an integrated PET-CT scanner located at Princess Margaret Cancer Centre.

The purpose of this study is to find out if the use of 68Ga-PNT6555 (FAPI) PET-CT will improve the assessment of disease extent as compared to routine CT scans. The radiopharmaceutical ("radiotracer") 68Ga-PNT6555 (FAPI) is experimental. Experimental means Health Canada has not approved the sale or use of 68Ga-PNT6555 (FAPI), but they have approved its use in this research study.

About 30 patients will take part in this study, and estimate it will take up to 3 years to complete the study enrollment.

Our primary goal is to determine if high-grade epithelial ovarian cancers have a strong affinity for 68Ga-PNT6555, which is a Fibroblast activation protein inhibitor also known as FAPI.

Our secondary objectives: Compare Positron Emission Tomography (PET) scan to CT (computerized tomography) and surgical findings, check FAPI uptake after chemotherapy and assess 68Ga-PNT6555 safety.

The Tertiary objectives aim to achieve are to detect residual disease with FAPI PET after primary cytoreduction, assess expression variation at different tumour sites, and determine correlations between FAP tumour volumes and clinical parameters such as cytoreduction, Progression-free survival (PFS), and overall survival (OS).

This study focuses on individuals who have been diagnosed or are suspected to have high-grade serous ovarian cancers (HGSOC). They must have had a CT scan of their abdomen and pelvis within 6 weeks before enrolling in the study and be at clinical stage III or IV. These individuals must also be considered for primary cytoreductive surgery or neoadjuvant chemotherapy. During the study, patients will undergo a PET/CT scan at the outset and a follow-up scan within six weeks of the screening.

For those who are receiving chemotherapy and then interval cytoreductive surgery, additional scans will be scheduled. Patients who have undergone complete cytoreduction can arrange a scan four weeks after the surgery.

In order to participate in this study, certain criteria must be met. These include being at least 18 years of age, having received a diagnosis of HGSOC via cytology or histology, or having clinical suspicion of HGSOC based on various factors such as symptoms, physical exam, tumour markers, and imaging findings. It is also necessary to have clinical stage III or IV, be considered for primary Cytoreductive Surgery(PCS)or NACT, and have had a contrast-enhanced CT abdomen and pelvis within 6 weeks of PET prior to enrolling. Informed consent and adherence to PET examination safety guidelines are required for participation in this study. Eligibility criteria include the absence of pregnancy, the ability to remain still during the exam, and the absence of certain types of ovarian cancer or advanced gynecological malignancy, such as mucinous, low-grade serous, low-grade endometrioid, and low-malignant potential tumours. Throughout the procedure, patients who are receiving 68Ga-PNT6555 will be injected with a precisely measured dose of 120-220 MBq(Mega Becquerel - Unit of activity of a quantity of radioactive material)(3.2-5.9 mCi) via a syringe over a period of 5-10 seconds. Following that, they will undergo a 60-120-minute uptake time and are required to drink 750 mL of dilute water-soluble oral contrast, which is a standard protocol for PET/CT in abdominal malignancies. A low-dose CT scan will be obtained from mid-skull to mid-thigh, followed by 3D PET acquisition. Attenuation correction and emission reconstruction will be carried out according to standard clinical practices. The scan parameters will be meticulously documented in accordance with departmental guidelines. Patient safety will be closely monitored throughout the scanning session and up to 2 hours after the radiopharmaceutical injection. Prior to taking part in the research, all potential candidates will undergo a thorough screening process to verify their eligibility. Following this, they will sign an Informed Consent Form and the Clinical research Coordinator( CRC) will complete a registration checklist. The PI will closely oversee the clinical research coordinator's management of data and record keeping to guarantee that they are precise, comprehensive, easy to read, and punctual. Based on the limited clinical experience with 68Ga-PNT6555, the risk of significant side effects is low. Available information indicates that over 100 patients who received a similar dye reported no side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion in this study if they meet the following criteria:

  * Age ≥18 years.
  * Cytological or histological diagnosis of HGSOC, or clinical suspicion of HGSOC based on symptoms, physical exam, tumour markers, and imaging findings.
  * Clinical stage III or IV, being considered for PCS or NACT.
  * Contrast-enhanced CT abdomen and pelvis within 6 weeks of PET (prior to enrolment).

Exclusion Criteria:

Patients will be ineligible to participate in this study if they meet any of the following criteria:

* Inability to provide informed consent.
* Contraindications for PET examination as per institutional safety guidelines, including but not limited to pregnancy, or inability to lie still for PET examination.
* Evidence of the following epithelial ovarian cancer histological subtypes: Mucinous, low-grade serous, low-grade endometrioid, and low-malignant potential tumours.
* Non-ovarian advanced gynecological malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — individuals who have been diagnosed or are suspected to have high-grade serous ovarian cancers (HGSOC).
Enrollment: 30 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
FAPI positivity | through study completion, an average of 1 year
  A lesion will be considered abnormal when focal tracer accumulation is greater than background activity and cannot be attributed to a physiological or benign entity.FAPI tumour volumes will be correlated with clinical outcome measures including:
  1. Achievement of optimal or complete cytoreduction;
  2. Progression-free survival (PFS);
  3. Overall survival (OS).
Quantitative parameters | through study completion, an average of 1 year
  Comparison of tracer uptake (SUVmax/mean) in a lesion to reference tissues (blood pool, liver); calculation of ratio of lesion SUV/ reference tissues.

SECONDARY OUTCOMES:
Modality performance measures (CT vs PET) | through study completion, an average of 1 year
  Sensitivity, specificity, Negative Predictive Value (NPV), Positive Predictive Value (PPV) and validity will be calculated for each modality according to the reference standard (surgery and surgical histopathology) for all evaluable lesions.
Frequency of AE's | through study completion, an average of 1 year
  Safety Measurements

IPD SHARING:
Plan to Share IPD: No